CLINICAL TRIAL: NCT02434653
Title: A Comparison Between Two Strategies for Postpartum Anemia Diagnosis and Follow up After Vaginal Deliveries - Hemoglobin Screening in High Risk Population Versus by Symptoms
Brief Title: A Comparison Between Two Strategies for Postpartum Anemia Diagnosis and Follow up After Vaginal Deliveries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, enav yefet, MD/PhD, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0112-14
Record Dates: First submitted 2015-04-28; First posted 2015-05-05 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-05

CONDITIONS: Postpartum Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postpartum anemia diagnosis following symptoms (Experimental): Post partum anemia will be assessed by taking hemoglobin level following symptoms consistent with anemia, severe postpartum hemorrhage or hemoglobin level below 8 g/dL in the first 5 days following delivery
  Interventions: Other: Monitoring hemoglobin levels following anemia associated symptoms
- Postpartum anemia diagnosis following patients screening (Experimental): Post partum anemia will be assessed by taking hemoglobin level in patients at increased risk to develop post-partum anemia in the first 5 days following delivery, defined as patients with initial (before or immediately after delivery) hemoglobin level of 10.5 g/dl or less regardless of symptoms, or in cases of severe post partum hemorrhage.
  Interventions: Other: Monitoring hemoglobin levels to detect anemia by screening of women at increased risk for post partum anemia

INTERVENTIONS:
Other: Monitoring hemoglobin levels following anemia associated symptoms — Post-partum anemia will be diagnosed after vaginal delivery by taking hemoglobin levels to patients with symptoms consistent with anemia, severe postpartum hemorrhage or hemoglobin level below 8 g/dL.
  Arms: Postpartum anemia diagnosis following symptoms
Other: Monitoring hemoglobin levels to detect anemia by screening of women at increased risk for post partum anemia — Post-partum anemia will be diagnosed after vaginal delivery by taking hemoglobin levels to high risk women for post-partum anemia, defined as hemoglobin levels of 10.5 g/dl or below around delivery, or severe postpartum hemorrhage with or without symptoms associated with anemia
  Arms: Postpartum anemia diagnosis following patients screening

SUMMARY:
Anemia diagnosis by hemoglobin level monitoring in women after vaginal delivery by symptoms versus screening of women at increased risk for post-partum anemia.

DETAILED DESCRIPTION:
Anemia is common following delivery. It is associated with some serious complications including increased risk for syncope and in severe cases even cardiogenic shock. Yet, anemia-associated symptoms might manifest relatively late after the patient have lost a fair amount of blood, which was not diagnosed early enough. To date, there are not acceptable guidelines for monitoring hemoglobin levels after delivery. Theoretically, there are 2 approaches for hemoglobin monitoring - one by taking hemoglobin levels in order to diagnose anemia in patients reporting anemia-associated symptoms. The other approach is by screening of women at increased risk for post-partum anemia. In the present study we aimed to compare those 2 approaches.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women after vaginal delivery

Exclusion Criteria:

* pregnant women with known sensitivity to the product iron sucrose
* pregnant women after cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1679 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The rate of patients diagnosed with anemia | Up to 3 days postpartum
  Hemoglobin of 10 g/dl or below
The rate of patients who received treatment with intravenous iron sucrose | Up to 3 days postpartum

SECONDARY OUTCOMES:
The rate of patients who received blood transfusion | From delivery and up to 5 days
The rate of women with post-partum hemorrhage | From delivery and up to 5 days
The rate of women who underwent uterine revision following delivery after their arrival to the maternity ward | From delivery and up to 5 days
The rate of women who needed uterotonic agents after their arrival to the maternity ward | From delivery and up to 5 days
The average blood tests number that was performed | From delivery and up to 5 days
Minimal and average hemoglobin level | From delivery and up to 5 days
The composite symptoms of anemia and functional capacity after 6 weeks postpartum as assessed by a questionnaire | 6 weeks postpartum
  Each question in the questionnaire will receive a score. The total score will be reported.
Hemoglobin level 6 weeks postpartum | 6 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek Medical Center, Afula, Israel

REFERENCES:
- [Derived] Yefet E, Yossef A, Nachum Z. Prediction of anemia at delivery. Sci Rep. 2021 Mar 18;11(1):6309. doi: 10.1038/s41598-021-85622-7. PMID 33737646